# Combined Document: Study Protocol, Statistical Analysis Plan (SAP), and Informed Consent Form (ICF)

Official Title of the study: Behavioral change communication intervention in menstrual disorder management among female university students in Bangladesh

Professor Dr. GM Rabiul Islam

Principal investigator of the study

Shahjalal University of Science and Technology (SUST), Sylhet, Bangladesh

Document date: 26 May 2025

Approved by the SUST Research Ethics Board (Ref: AST/002/258)

# **Study Protocol**

# **Brief summery**

Menstrual health is a neglected area of women's health research, especially in low- and middle-income countries, despite the high prevalence and impact of menstrual disorders on daily life. These issues are particularly common among young women in academic settings, yet few interventions address them holistically. In Bangladesh, female university students frequently experience dysmenorrhea, premenstrual syndrome (PMS), and menstrual irregularity (MI), conditions often worsened by modifiable lifestyle factors such as poor diet, physical inactivity, and food cravings. This study assessed the effectiveness of Behavior Change Communication (BCC) intervention promoting non-pharmacological strategies to improve menstrual health among female university students.

A quasi-experimental design included 498 participants (249 per group), aged 19–25, from three public universities. The intervention group received three interactive BCC sessions on menstrual disorders, diet, and physical activity (including yoga) between May and June 2023, followed by bi-monthly visits for six months. Post-intervention data were collected from February to March 2024. Outcomes (dysmenorrhea, PMS, MI) were measured using validated tools. Propensity score matching (1:1 nearest-neighbor, caliper = 0.01) yielded 98 matched participants per group. Covariates included physical activity, body mass index (BMI), dietary diversity, food cravings, breakfast skipping, sleep, bedtime, caffeine intake, and socio-demographic factors. Data were collected via validated Bengali questionnaires. Analyses included descriptive statistics, chi-square and t-tests, logistic regression, and sensitivity analyses. Ethical approval was granted by the Shahialal University Ethics Board.

# **Detailed description of the study**

Menstrual health is a significantly under-researched aspect of women's health, particularly among adolescents and young adults in low- and middle-income countries(1), even though menstrual disorders affect up to 75% of them and often interfere with daily functioning and overall well-being. (2). In Bangladesh, female university students frequently experience menstrual disorders such as dysmenorrhea, premenstrual syndrome (PMS), and menstrual irregularity (MI). These conditions are often aggravated by modifiable lifestyle factors including poor dietary intake, physical inactivity and food cravings for high fat and sweet food (3).

This study evaluated the effectiveness of a structured behavior change communication (BCC) intervention designed to improve menstrual health among female university students in Bangladesh. The intervention focused on three key menstrual health outcomes: dysmenorrhea, PMS, and MI. It promote a sustainable, non-pharmacological approach to managing common menstrual disorders through behavior and lifestyle changes including improved physical activity and dietary diversity.

The study employed a quasi-experimental design involved two groups: an intervention group that received BCC module and a control group that did not. Participants were female undergraduate students aged 19 to 25 years, residing in dormitories at three public universities in Bangladesh i.e. Patuakhali Science and Technology University (PSTU), Barishal University (BU), and Khulna University (KU). Ethical approval was obtained from the Shahjalal University of Science and Technology Research Ethics Board (Ref. No. AST/002/258), and all participants provided written informed consent. The BCC intervention comprised three interactive educational sessions

delivered between May 20 and June 30, 2023, by trained female facilitators. The first session addressed menstrual disorders and associated risk factors, the second focused on healthy dietary practices, and the third emphasized physical activity (including yoga) and other relevant lifestyle modifications. To reinforce the content, follow-up visits were conducted every two months over a six-month period. Post-intervention data collection was carried out between February and March 2024.

A total of 498 participants (249 in each group) were initially enrolled, based on power calculations designed to detect a 30% reduction in the prevalence of menstrual disorders, with 80% statistical power and 95% confidence level. After exclusions for missing data and loss to follow-up, 234 intervention and 238 control participants were included in the analysis of dysmenorrhea; and 228 participants per group were retained for PMS and MI outcomes. To reduce selection bias and ensure covariate balance, 1:1 nearest-neighbor propensity score matching (PSM) was applied using a logistic regression model with a caliper of 0.01 and no replacement. The final matched sample included 196 participants (98 per group) for each outcome.

Among all the primary outcomes, dysmenorrhea was assessed using the Andersch and Milsom (4) four-point scale and dichotomized as no pain (Grade 0) vs. any pain (Grades 1-3). PMS was evaluated by the premenstrual symptoms screening tool (PSST) and recoded into a binary variable: No/Mild PMS (code = 0) and Moderate to Severe PMS or premenstrual dysphoric disorder (PMDD) (code = 1) (5). Additionally, Menstrual irregularity was determined based on self-reported cycle length and coded as irregular (1) if <21 or >35 days, and not irregular (0) if within the 21-35 day range (6).

The treatment variable was exposure to the BCC intervention (yes/no). The covariates included physical activity, obesity, dietary habits, lifestyle factors, and socio-demographic characteristics. Physical activity was classified according to WHO guidelines (7) as: (i) sedentary: light-intensity activities; (ii) active: moderate-intensity activities for 150–300 minutes per week; and (iii) athlete: vigorous-intensity activities for 75–150 minutes per week. Obesity was assessed using body mass index (BMI, kg/m²) and categorized according to WHO Asian-specific cut-offs (8): (i) underweight (<18.5), (ii) normal weight (18.5–22.9), (iii) overweight (23.0–27.5), and (iv) obese (>27.5). Dietary information was collected using a five-day 24-hour recall method, and dietary diversity score (DDS) was calculated following FAO guidelines (9). Lifestyle-related covariates included food cravings for high-fat or sweet foods (10), skipping breakfast, sleep duration, bedtime and caffeine intake (11). Socio-demographic variables included family history of menstrual disorders, age at menarche, marital status, and participants' residence as well as parental educational and occupational status.

Data were collected through interviewer-administered, culturally adapted, and validated Bengali-questionnaires. Descriptive statistics summarized baseline characteristics. Group differences were tested using chi-square and t-tests. Propensity scores were estimated using logistic regression, and covariate balance post-matching was evaluated using standardized mean differences (SMD <10%). Intervention effects were analyzed using conditional logistic regression on the matched sample, and logistic regression (bivariate/multivariate) on the unmatched sample. Sensitivity analyses included covariate balance diagnostics, estimation of average treatment effects (ATE/ATT), and Bayesian logistic regression with log Bayes factor.

This study complies with U.S. regulatory requirements for clinical trial registration and reporting under 42 CFR Part 11. The responsible party confirms that all submitted information is complete and accurate, and that the study protocol, statistical analysis plan (SAP), and informed consent form (ICF) reflect the approved trial objectives and design.

# Participant flow

#### **Recruitment details**

Female students were recruited from three public universities in Bangladesh: Patuakhali Science and Technology University (PSTU), Barisal University (BU), and Khulna University (KU) for a BCC module on menstrual health from May 20 to June 30, 2023. Recruitment occurred via campus outreach and voluntary registration. University-approved session dates were held in campus venues. Follow-up occurred from July 15, 2023, to January 15, 2024. A post-intervention assessment was conducted from February to March 2024 through comparing the intervention group to the control group.

## **Pre-assignment details**

Initially 498 participants (249/group) were recruited. Seven intervention participants were excluded before assignment for missing sessions/protocol violation, leaving 242. At six-month follow-up, 480 participants (239 intervention, 241 control) completed assessments as because 3 intervention and 8 control participants were excluded due to missed follow-up or withdrawal. After data checks, 8 were excluded for invalid dysmenorrhea data, leaving 234 intervention and 238 control (total 472 participants) for that outcome. For PMS and MI, 24 more were excluded (10

intervention and 14 control group), yielding 456 participants (228 per group). Propensity score matching (PSM) identified 196 matched participants (98 per group) for each of outcomes.

## **Group information**

Two groups were assigned: an intervention group receiving the BCC module on menstrual health, and a control group with no intervention. Participants were female university students from PSTU, BU, and KU, Bangladesh, with group assignment based on attending at the BCC sessions.

#### **Group title**

- 1. Intervention Group
- 2. Control Group

#### **Group description**

The Intervention group comprised female university students from PSTU, BU, and KU who participated in a structured BCC module designed to enhance awareness and promote effective management of menstrual disorders through lifestyle and behavioral modifications. The module consisted of three interactive sessions that included educational presentations, yoga demonstrations, informational pamphlet distribution, quiz competitions, and small gift incentives to boost engagement. Sessions were facilitated by trained female educators under the guidance of a public health expert and a gynecologist. Participants were selected through voluntary registration and received follow-up support at every two months to reinforce behavioral changes, address challenges, and ensure continued adherence to healthy practices.

The Control group consisted of female students from the same universities who were not exposed to the BCC intervention. They were selected using student dormitory records and matched to the intervention group through propensity score matching to ensure comparability. As they did not receive any form of menstrual health education or BCC intervention, this group served as the baseline comparator for evaluating the effectiveness of the BCC module on menstrual health outcomes.

#### Period(s)

This study was organized into three distinct periods to reflect the logical progression of the intervention and its evaluation: (1) implementation of the intervention, (2) follow-up phase to monitor and support behavior change, and (3) post-intervention evaluation to assess outcomes. Each period captured critical milestones and participant flow to assess the feasibility, adherence, and effectiveness of the intervention.

#### **Period 1: Implementation of the intervention**

The first period of the study involved the implementation of a structured BCC intervention among female university students to enhance awareness and promote effective management of menstrual disorders. Three structured sessions were conducted covering menstrual disorders, dietary behaviors, and physical activity. Two trained female educators facilitated these sessions. The details of participation status of this period is presented in Table 1.

Table 1. Summary of participation status and key milestones in intervention implementation

| Participation status | Data<br>(number of<br>participants) | Comments | Milestone title | Milestone data (number of participants) |
|---|---|---|---|---|
| Started | 249 (Intervention Group) 249 (Control group) | Intervention: participants who registered after informed consent and attended the first session of BCC module Control: Participant from the same universities were | Intervention: first session attendance Control: Not exposed to the | 249 (Intervention Group) 249 (Control |
| | | selected and listed after providing consent for the assessment study. | BCC intervention | group) |
| Completed | 242 (Intervention Group) | Participants who attended all three intervention sessions. | Completed all sessions | 242 |
| Not completed | 7<br>(Intervention Group) | Participants dropped out<br>before completing the 2nd<br>and/or 3rd session. | Protocol violation | 7 |

## **Period 2: Follow-up phase**

This was a six-month post-intervention follow-up period, during which participants in the intervention group received periodic support visits to reinforce behavioral changes and sustain the practices introduced during the BCC sessions (Table 2).

Table 2. Overview of participation status and milestone achievements in follow-up phase

| Participation status | Data<br>(number of<br>participants) | Comments | Milestone title | Milestone<br>data<br>(number of<br>participants) |
|---|---|---|---|---|
| Started | 242<br>(Intervention Group) | Participants who completed all the sessions of the intervention and entered follow-up phase. | Follow-up initiated and available at first follow-up visit | 242 |

| Completed | 239 | Participants available at 6- | Follow-up | 239 |
|---|---|---|---|---|
| | (Intervention Group) | month follow-up assessment. | completed | 239 |
| Not completed | 3 (Intervention Group) | Participants lost to follow-up during the periodic monitoring visits conducted every two months. | Lost to follow-up | 3 |

#### **Period 3: Post-intervention evaluation**

This period represents the final stage of the study to assess the effectiveness of the BCC module on key menstrual health outcomes through a quasi-experimental design using matched control and intervention participants (1:1 PSM) (Table 3, Table 4A and 4B). Outcome assessments were done for dysmenorrhea, PMS and MI.

Table 3. Participant flow and milestone completion in post-intervention outcome evaluation before matching

| Participation status | Outcomes | Data<br>(number of<br>participants) | Comments | Milestone<br>title | Milestone<br>data<br>(number of<br>participants) |
|---|---|---|---|---|---|
| Started | Dysmenorrhea,<br>PMS and MI | 239 (Intervention),<br>241 (Control) | Participants agreed to join and assessed for final evaluation of outcomes | Assessment initiated | 480 |
| Completed | Dysmenorrhea | 234 (Intervention),<br>238 (Control) | Participants included after cleaning for dysmenorrhea outcomes. | Valid responses | 472 |
| Completed | PMS and MI | 228 (Intervention),<br>228 (Control) | Final sample included participants with valid PMS and IMC outcome data | Appropriate responses | 456 |
| Not completed | Dysmenorrhea | 8 (5 intervention and 3 control) | Omitted from the final dataset due to | Incomplete response | 8 |

| | | data quality issues,<br>including missing or<br>invalid responses | | |
|---|---|---|---|---|
| PMS and MI | 24 (11 intervention and 13 control) | Removed from analysis because of incomplete or inaccurate data. | Invalid<br>response/<br>missed data | 24 |

Table 4A. Participation flow of matched sample for post-intervention dysmenorrhea analysis

| Participation status | Groups | Data<br>(number of<br>participants) | Comments | Milestone<br>title | Milestone<br>data<br>(number of<br>participants) |
|---|---|---|---|---|---|
| Started | Intervention | 234 | Out of 234 eligible participants, 98 were selected using PSM and individually matched in a 1:1 ratio with control participants within the common support region. | Enrollment | 472 |
| | Control | 238 | All participants initially eligible; matched pool was drawn from this group | | |
| | Intervention | 98 | All 98 matched completed the post-intervention evaluation | Matching | |
| Completed | Control | 98 | 98 matched controls completed the evaluation and the remaining controls not matched due to 1:1, noreplacement rule | completion<br>and final<br>outcome<br>analysis | 196 |
| Not completed | Intervention | 136 | The participants were excluded from the analysis because they could not be matched with any control participants within the specified caliper of 0.01 | Excluded due to fall outside the region of common support | 276 |
| Not completed | Control | 140 | Even though these participants fell within the common support region, they were excluded because of the 1:1 matching requirement and the no-replacement rule. | Not selected<br>due to 1:1<br>matching<br>without<br>replacement | |

Table 4B. Matched sample of participants for post-intervention assessment of PMS and MI outcomes

| Participation status | Groups | Data<br>(number of<br>participants) | Comments | Milestone<br>title | Milestone<br>data<br>(number of<br>participants) |
|---|---|---|---|---|---|
| Started | Intervention | 228 | From the pool of 228 eligible participants, 98 were chosen using PSM and matched one-to-one with control participants within the common support region. A subset of matched | Enrollment | |
| | Control | 228 | participants was selected from all 228 initially eligible control individuals | | 456 |
| Completed | Intervention | 98 | All 98 participants in the matched group successfully completed the post-intervention assessment. | Matching completion | |
| | Control | 98 | The evaluation was completed<br>by 98 matched control<br>participants while the rest were<br>excluded in accordance with<br>the 1:1 matching and no-<br>replacement criteria. | and final<br>outcome<br>analysis | 196 |
| Not completed | Intervention | 130 | As no matches within the caliper of 0.01 could be identified, the participants were excluded from the analysis | Participants were excluded as they did not fall within the region of common support. | 260 |
| | Control | 130 | Despite being within the common support region, these participants were excluded to maintain the 1:1 matching ratio and adhere to the noreplacement rule. | Excluded because of 1:1 matching without replacement. | |

## **Baseline characteristics**

## **Group information**

#### **Group title**

- 1. Intervention Group
- 2. Control Group

#### **Group description**

The intervention group included participants who attended all three sessions of the BCC module on menstrual health management. Initially, 249 participants were recruited, and 242 completed all sessions. At the six-month follow-up, 239 participants completed the outcome assessment. After data cleaning, 234 participants were eligible for the final analysis of the dysmenorrhea outcome, while 228 participants had valid data and were included in the analyses of PMS and MI.

Participants in the control group did not receive the BCC intervention but were matched in number and characteristics to the intervention group. Initially, 249 participants were listed for the control arm, and 241 completed the outcome assessment interview. Following data quality verification, 238 participants were included in the final analysis for the dysmenorrhea outcome. For the PMS and MI outcomes, 228 participants had valid and complete data and were included in the respective analyses.

After propensity score matching, 98 matched participants from each group (n=196) were used for the final analysis of each outcome variable, ensuring balance between the groups on key covariates.

## **Baseline analysis population information**

The baseline analysis populations differ slightly from the initial recruitment numbers due to participant withdrawal, non-response, absence during sessions or protocol violation, and exclusion based on data quality checks for outcome variables (Table 5).

Table 5. Baseline Profile of Participants by Study Group: Intervention vs. Control

| Outcome | Group | Overall number<br>of baseline<br>participants | Baseline analysis population description |
|---|---|---|---|
| | Intervention | 234 | After recruitment and data quality checks, 234 participants were included in the initial analysis. After propensity score matching, 98 were retained. |
| Dysmenorrhea | Control | 238 | From 238 eligible controls, 98 matched participants were used in the final matched analysis. |
| | Total | 472 | The final matched sample included 196 participants (98 per group), selected through 1:1 propensity score matching without replacement using a caliper of 0.01. |
| | Intervention | 228 | 228 participants provided valid and complete responses and were included in the baseline analysis. After matching, 98 were included in the final matched analysis. |
| PMS and MI | Control | 228 | 228 participants were eligible for baseline analysis. After matching, 98 were used for final analysis. |
| | Total | 456 | A total of 196 participants (98 in each group) were retained after 1:1 matching with a 0.01 caliper and no replacement. |

#### **Baseline Measure Information**

The baseline characteristics of study participants were assessed using a combination of study-specific and standard measures to comprehensively capture their lifestyle, nutritional, reproductive, and socio-demographic profiles (Table 6). Study-specific measures included

physical activity level (categorized according to WHO guidelines), body mass index (BMI) using Asian-specific cut-offs, and minimum dietary diversity (MDD) based on a 5-day food diary aligned with FAO recommendations. Additional lifestyle factors assessed included food cravings, skipping breakfast, sleep duration, caffeine intake frequency, and bedtime. Reproductive health and demographic factors such as age, age at menarche, marital status, and participant's residence, family history of menstrual disorders, as well as parental education and occupation were also recorded. These baseline measures were used to describe the participant population and to adjust for potential confounding in subsequent analyses.

To evaluate the impact of the BCC intervention on reducing dysmenorrhea, key covariates were balanced between groups using propensity score matching. These included physical activity level, BMI, minimum dietary diversity (MDD score  $\geq 5$ ), food cravings for high-fat and sweet foods, breakfast skipping, sleep duration, caffeine intake frequency, family history of menstrual disorders, age at menarche, marital status, father's and mother's educational status, and mother's occupation. These balanced covariates (13 covariates) were included in the regression models and in the estimation of both the average treatment effect (ATE) and the average treatment effect on the treated (ATT).

Additionally, to assess the effectiveness of the intervention on PMS and MI outcomes, propensity score matching was used to achieve balance in key baseline covariates between the intervention and control groups. The matched covariates included physical activity level, BMI ( $kg/m^2$ ), minimum dietary diversity (MDD score  $\geq 5$ ), food cravings for high-fat and sweet foods, breakfast skipping, sleep duration, age at menarche, and participants' residence. These variables (8 covariates) were subsequently adjusted for in the estimation of treatment effects.

Table 6. Baseline characteristics of participants by defined study measures

| Baseline<br>measure title<br>(Study-specific<br>measure) | Study-specific<br>baseline measure<br>title(s) | Baseline measure description | Measure<br>type | Measure<br>of<br>dispersion | Category<br>title | Unit of measure |
|---|---|---|---|---|---|---|
| Physical activity | Physical activity level | Categorized per WHO recommendations based on weekly activity intensity: sedentary (with little or no activity), active (moderate, 150–300 min/week) and athlete (vigorous, 75–150 min/week). Active and athlete were merged during analysis | Count of participants | Not<br>applicable | Sedentary/<br>Active and<br>athlete | Participants |
| Body mass index (BMI) | BMI (Kg/m²) | Classified using WHO cut-offs for Asian populations, such as underweight (<18.5), normal (18.5–22.9) and overweight/obese (≥23.0). Overweight and obese categories were merged. | Count of Participants | Not applicable | Underweight /<br>Normal /<br>Overweight<br>and obese | Participants |
| Dietary diversity<br>Score (DDS) | MDD (scoring ≥ 5) | Dietary diversity was assessed using a 5-day food diary based on the 24-hour recall method, following FAO guidelines. Food items were classified into 10 predefined groups, and scores ranged from 0 to 10. Minimum dietary diversity (MDD) was defined as achieving a score of 5 or more. | Count of participants | Not<br>applicable | Yes / No | Participants |
| Food Craving | Food craving for high-fat and sweet food | Self-reported craving for high-fat and sweet food. | Count of participants | Not applicable | Yes / No | Participants |
| Skipping<br>breakfast | Skipping breakfast | Reported skipping breakfast one or more times during the last week. | Count of participants | Not applicable | Yes / No | Participants |
| Sleep duration | Sleep hours per night | Based on self-reported average nightly sleep duration | Count of participants | Not applicable | <7 hrs /≥7 hrs | Participants |
| Caffeine consumption | Frequency of caffeine Intake | Based on frequency of caffeine intake per week; categorized as infrequent (<3 times/week) or frequent (≥3 times/week) | Count of participants | Not applicable | Infrequent / Frequent | Participants |

| Bedtime | Bedtime (hours) | Bedtime was classified into two groups:<br>≤23:00 hours and >23:00 hours, based on a<br>24-hour clock format | Count of participants | Not applicable | Before or at 23:00 / After 23:00 | Participants |
|---|---|---|---|---|---|---|
| Family history of menstrual disorders | Family history of menstrual disorders | Participants reported whether they had family history of any kind of menstrual disorders viz. dysmenorrhea, PMS, or IMC. | Count of participants | Not applicable | Yes / No | Participants |
| Age (Not study- specific measure) | Age | Treated as continuous variable | Mean | Standard deviation | Not applicable | Participants |
| Menarche age | Age at menarche | Reported age at first menstruation in years and treated as continuous variable. | Mean | Standard deviation | Not applicable | Participants |
| Marital status | Marital status | Marital status was self-reported. Participants categorized as divorced, separated, or recently married were grouped under ever married. All others were classified as never married. | Count of participants | Not applicable | Never married<br>/ Ever married | Years |
| Residence | Participant's residence | Living arrangement of the participants during the study time. | Count of participants | Not applicable | With Family /<br>at student<br>dormitory | Participants |
| Father's<br>Education | Father's educational status | Education levels were categorized as: "Below secondary education" (no formal education, primary, or incomplete secondary schooling) and "Secondary or higher | Count of participants | Not applicable | Below<br>Secondary (0-<br>5 y schooling)<br>/ Secondary | Participants |
| Mother's<br>Education | Mother's educational status | education" (completed secondary school, higher secondary, college, or university) | | | and above(> 5 y schooling) | |
| Father's Occupation Mother's Occupation | Father's occupational status Mother's occupational status | Occupational status was self-reported as either Formal (salaried or secure jobs) or Informal (homemaking, daily wage, or insecure work) | Count of participants | Not applicable | Formal /<br>Informal | Participants |

#### **Number of baseline participants**

The number of baseline participants is the same as the overall number of baseline participants, as it includes all individuals who completed baseline data collection and met the data quality criteria. Although PSM was later used to create comparable groups for outcome analysis, the baseline measures reflect the entire recruited sample before matching. Therefore, no separate or reduced sample size is reported in this section.

#### **Baseline Measure Data**

Baseline characteristics were assessed at the time of outcome evaluation for both the intervention and control groups. Although data were collected post-intervention, propensity score matching was applied to balance pre-existing covariates and reduce selection bias in estimating the treatment effect. The Table 7(A and B) present the baseline values for each measure across the intervention and control groups, as well as for the total study population.

Table 7A. Comparison of baseline characteristics between study groups for dysmenorrhea outcome

| Variables | Control | Intervention | Total |
|---|---|---|---|
| Variables | (n = 238) | (n = 234) | (N=472) |
| Physical activity level | | | |
| Sedentary | 206 (43.6) | 114 (24.2) | 320 (67.8) |
| Active and Athlete | 32 (6.6) | 120 (25.6) | 152 (32.2) |
| $BMI(kg/m^2)$ | | | |
| Normal weight (18.5-22.9) | 83 (17.6) | 171 (36.2) | 254 (53.8) |
| Underweight (<18.5) | 44 (9.3) | 37 (7.8) | 81 (17.2) |
| Overweight and obese (>22.9) | 111 (23.5) | 26 (5.5) | 137 (29.0) |
| $MDD$ (scoring $\geq 5$ ) | | | |
| No | 153 (32.4) | 96 (20.3) | 249 (52.8) |
| Yes | 85 (18.01) | 138 (29.2) | 223 (47.2) |
| Food craving for high fat and sweet food | | | |
| No | 77 (16.3) | 164 (34.8) | 241 (51.1) |

| Yes | 161 (34.1) | 70 (14.8) | 231 (48.9) |
|---------------------------------------|------------|------------|------------|
| Skipping breakfast | <u> </u> | <u> </u> | |
| No | 72 (15.5) | 169 (35.8) | 241 (51.1) |
| Yes | 166 (35.2) | 65 (13.8) | 231 (48.9) |
| Sleep hours per night | | | |
| ≥7 hours | 75 (15.9) | 155 (32.8) | 230 (48.7) |
| < 7 hours | 163 (34.5) | 79 (16.7) | 242 (51.3) |
| Frequency of caffeine Intake | l | l | |
| Infrequent (< 3 times per week) | 65 (13.8) | 157 (33.3) | 222 (47.0) |
| Frequent $\geq 3$ times per week) | 173 (36.7) | 77 (16.3) | 250 (53.0) |
| Bedtime (hours) | l | l | |
| Before or at 23:00 | 26 (5.5) | 139 (29.5) | 165 (35.0) |
| After 23:00 | 212 (44.9) | 95 (20.1) | 307 (65.0) |
| Family history of menstrual disorders | <u> </u> | 1 | |
| No | 160 (33.9) | 197 (41.7) | 357 (75.6) |
| Yes | 78 (16.5) | 37 (7.8) | 115 (24.4) |
| Age (years) | <u> </u> | 1 | |
| Mean (SD) | 21.9 (1.4) | 21.0 (1.5) | 21.5 (1.5) |
| Age at menarche (years) | • | 1 | |
| Mean (SD) | 12.1 (1.5) | 13.4 (1.7) | 12.7 (1.7) |
| Marital status | <u>.</u> | <u> </u> | |
| Never Married | 216 (45.8) | 226 (47.9) | 442 (93.6) |
| Ever married | 22 (4.7) | 8 (1.7) | 30 (6.4) |
| Place of residence | <u>.</u> | <u> </u> | |
| With Family | 18 (3.8) | 46 (9.8) | 64 (13.6) |
| At student dormitory | 220 (46.6) | 188 (39.8) | 408 (86.4) |
| Father's educational status | | • | |
| Secondary and above (> 5 y schooling) | 188 (39.9) | 217 (46.0) | 405 (85.8) |
| Below secondary (0-5 y schooling) | 50 (10.6) | 17 (3.6) | 67 (14.2) |
| Mother's educational status | <u>.</u> | <u> </u> | |
| Secondary and above (>5 y schooling) | 176 (37.3) | 195 (41.3) | 371 (78.6) |
| Below secondary (0-5 y schooling) | 62 (13.1) | 39 (8.3) | 101 (21.4) |
| Father's occupational status | <u>.</u> | <u>.</u> | |
| Formal occupation | 138 (29.2) | 144 (30.5) | 282 (59.8) |
| Informal occupation | 100 (21.2) | 90 (19.0) | 190 (40.2) |
| Mother's occupational status | | <u>.</u> | |
| Formal occupation | 66 (14.0) | 44 (9.3) | 110 (23.3) |
| Informal occupation | 172 (36.4) | 190 (40.3) | 362 (76.7) |

Table 7B. Distribution of baseline characteristics among intervention and control groups for PMS and MI outcomes

| | Control | Intervention | Total |
|---|---|---|---|
| Variables | (n = 228) | (n = 228) | (N = 456) |
| Physical activity level | | | |
| Sedentary | 197 (43.3) | 112 (24.6) | 309 (67.8) |
| Active and Athlete | 31 (6.8) | 116 (25.4) | 147 (32.2) |
| $BMI(kg/m^2)$ | <u>'</u> | <b>'</b> | |
| Normal weight (18.5 – 22.9) | 80 (17.5) | 167 (36.6) | 247 (54.2) |
| Underweight (< 18.5) | 42 (9.2) | 37 (8.1) | 79 (17.3) |
| Overweight/obese (> 22.9) | 106 (23.2) | 24 (5.2) | 130 (28.5) |
| $MDD$ (scoring $\geq 5$ ) | | | |
| No | 145 (31.8) | 93 (20.4) | 238 (52.2) |
| Yes | 83 (18.2) | 135 (29.6) | 218 (47.8) |
| Food craving for high fat and sweet food | | | |
| No | 75 (16.5) | 159 (34.9) | 234 (51.3) |
| Yes | 153 (33.5) | 69 (15.1) | 222 (48.7) |
| Skipping breakfast | | | |
| No | 67 (14.7) | 165 (36.0) | 232 (50.9) |
| Yes | 161 (35.3) | 63 (14.0) | 224 (49.1) |
| Sleep hours per night | | | |
| ≥ 7 hours | 71 (15.6) | 151 (33.1) | 222 (48.7) |
| < 7 hours | 157 (34.4) | 77 (16.9) | 234 (51.3) |
| Frequency of caffeine Intake | · | · | |
| Infrequent (< 3 times per week) | 60 (13.1) | 152 (33.3) | 212 (46.5) |
| Frequent (≥ 3 times per week) | 168 (36.9) | 76 (16.7) | 244 (53.5) |
| Bedtime (hours) | · | · | |
| 23:00 and before | 24 (5.3) | 137 (30.0) | 161 (35.3) |
| After 23:00 | 204 (44.7) | 91 (20.0) | 295 (64.7) |
| Family history of menstrual disorders | · | · | |
| No | 151 (33.1) | 191 (41.9) | 342 (75.0) |
| Yes | 77 (16.9) | 37 (8.1) | 114 (25.0) |
| Age (years) | · | · | |
| Mean (SD) | 22.0 (1.4) | 21.0 (1.5) | 21.5 (1.5) |
| Age at menarche (years) | · | · | |
| Mean (SD) | 12.2 (1.5) | 13.4 (1.7) | 12.8 (1.7) |
| Marital status | , | • | |
| Never Married | 206 (45.2) | 221 (48.5) | 427 (93.6) |
| Ever married | 22 (4.8) | 7 (1.5) | 29 (6.4) |
| Place of participant's residence | | | |

| With family | 17 (3.7) | 44 (9.87) | 61 (13.4) |
|---------------------------------------|------------|------------|------------|
| At student dormitory | 211 (46.3) | 184 (40.3) | 395 (86.6) |
| Father's educational status | | | |
| Secondary and above (> 5 y schooling) | 180 (39.5) | 212 (46.5) | 392 (86.0) |
| Below secondary (0 – 5 y schooling) | 48 (10.5) | 16 (3.5) | 64 (14.0) |
| Mother's educational status | | | |
| Secondary and above (> 5 y schooling) | 168 (36.8) | 191 (41.9) | 359 (78.7) |
| Below secondary (0 – 5 y schooling) | 60 (13.2) | 37 (8.1) | 97 (21.3) |
| Father's occupational status | | | |
| Formal occupation | 130 (28.5) | 142 (31.1) | 272 (59.6) |
| Informal occupation | 98 (21.5) | 86 (18.9) | 184 (40.4) |
| Mother's occupational status | | | |
| Formal occupation | 65 (14.3) | 44 (9.3) | 109 (23.9) |
| Informal occupation | 163 (35.7) | 185 (40.6) | 348 (76.1) |

## **Outcome measures**

#### **Outcome measure information**

In accordance with the study protocol, this section (Table 8) details the predefined primary outcomes used to evaluate intervention efficacy. The study focused on three key outcomes: dysmenorrhea, PMS and MI. Each was measured during the post-intervention period using standardized assessment tools. To support the study's quasi-experimental design and statistical analysis, all outcome variables were recoded as binary indicators.

Table 8. Summary of outcome measures information

| Data elements | Dysmenorrhea | Premenstrual Syndrome<br>(PMS) | Menstrual Irregularity (MI) |
|---|---|---|---|
| Outcome measure | Primary | Primary | Primary |
| type | | | |
| Outcome measure | Prevalence of | Prevalence of PMS | Prevalence of MI |
| title | Dysmenorrhea | | |
| Outcome measure | Assessed according to | Premenstrual symptoms were | Menstrual irregularity |
| description | Andersch and Milsom | assessed using premenstrual | was assessed based on |

| | 1 (0 1 0 0 111 | | |
|---|---|---|---|
| | scale (Grades $0-3$ ) which | symptoms screening tool | participants' self- |
| | evaluated the pain intensity | (PSST) and categorized into | reported cycle lengths. |
| and its impact on daily | | three groups: No/Mild PMS, | A cycle was considered |
| | activities. The scale of pain | Moderate to Severe PMS, and | irregular (coded 1 = |
| | intensity was recoded into | premenstrual dysphoric disorder | Yes) if it was shorter |
| | binary: $0 = No$ (no pain), 1 | (PMDD). For analysis, these | than 21 days or longer |
| | = Yes (any pain: | were combined into a binary | than 35 days. Cycles |
| | mild/moderate/severe). | variable: $0 = No/Mild PMS$ and | within the 21–35 day |
| | | 1 = Moderate to Severe PMS or | range were classified as |
| | | PMDD | not irregular (coded 0 = |
| | | | No) |
| Outcome messeum | Participants received three BCC sessions over approximately 6 weeks, followed by | | |
| Outcome measure | regular support to encourage behavior change for up to 6 months, with monitoring every | | |
| time frame | two months. Final outcomes were assessed about 8 months after enrollment. | | |
| Outcome measure | Count of participants | Count of participants | Count of participants |
| data type | | | |
| Measure of | Not applicable | Not applicable | Not applicable |
| dispersion/precision | Not applicable | Not applicable | Not applicable |
| | Yes (Dysmenorrhea = 1)/ | Yes (Moderate to Severe | Yes (MI = 1)/ |
| Category title | No (Dysmenorrhea = 0) | PMS/PMDD = 1)/ | No $(MI = 0)$ |
| | | No (No/mild PMS = 0) | |
| Unit of Measure | Participants | Participants | Participants |

## **Group information**

#### **Group title**

- 1. Intervention Group
- 2. Control Group

#### **Group description**

The intervention group comprised female university students who attended all BCC sessions conducted between May 20 and June 30, 2023, followed by a six-month monitoring period that included scheduled follow-ups every two months through January 15, 2024. The sessions focused on menstrual health education, dietary improvements, and physical activity. At the end of the

follow-up, 239 participants completed the outcome assessment. After data cleaning, 234 participants were included in the final analysis for dysmenorrhea, while 228 with valid and complete data were analyzed for PMS and MI outcomes.

Participants in the control group did not receive the BCC intervention or any related educational sessions but were matched with the intervention group based on number and baseline characteristics. Of the 249 participants initially enrolled in the control arm, 241 completed the outcome assessment interview. After data quality checks, 238 participants were retained for the final dysmenorrhea analysis. For the PMS and MI outcomes, 228 participants with complete and valid data were included in their respective analyses.

After propensity score matching, 98 matched participants from each group (n=196) were used for the final analysis of each outcome variable, ensuring balance between the groups on key covariates.

#### **Analysis population information**

This section provides (Table 9) an overview of the analysis populations for each outcome measure, including the number of participants at baseline and after propensity score matching. It also outlines the methods used to define the final samples included in the analyses.

Table 9. Overview of analysis population by groups for outcome measures

| Outcomes | Group | Overall number of participants analyzed | Analysis population description |
|---|---|---|---|
| | Intervention | 234 | Following initial recruitment and data quality verification, 234 participants in the intervention group and 238 in the |
| Dysmenorrhea | Control | 238 | control group were eligible for analysis. However, Final analyses were conducted using 1:1 propensity score |
| | Total | 472 | matching without replacement and a caliper of 0.01, yielding a matched sample of 196 participants (98 from each group). |
| | Intervention | 228 | For both PMS and IMC outcome measures, 228 participants from each group provided valid and complete |
| PMS and MI | Control | 228 | responses for the baseline analysis. Following 1:1 propensity score |
| | Total | 456 | matching without replacement (caliper = 0.01), 98 participants per group were retained, yielding a final matched sample of 196. |

#### Outcome measure data

Table 10 represents the outcome measure data for all participants who completed the follow-up assessment. Results are shown separately for the intervention and control groups, with each outcome reported as the number and percentage of participants. The data reflect the prevalence of each specified condition at follow-up, according to group assignment.

Table 10. Prevalence of key menstrual disorders among participants in control and intervention groups

| Outcome variables | Control (n = 238) | Intervention (n = 234) | Total (N = 472) |
|---|---|---|---|
| Prevalence of Dysmenorrhea | 1 | 1 | |
| No | 29 (6.1) | 159 (33.7) | 188 (39.8) |
| Yes | 209 (44.3) | 75 (15.9) | 284 (60.2) |
| | 1 | | |
| Outcome variables | Control | Intervention | Total |
| Outcome variables | (n = 228) | (n = 228) | (N = 456) |
| Prevalence of premenstrual syndrome (PMS) | · | · | |
| No/Mild PMS | 83 (18.2) | 205 (45.0) | 288 (63.2) |
| Moderate to Severe PMS/PMDD | 145 (31.8) | 23 (5.0) | 168 (36.8) |
| Prevalence of Menstrual Irregularity (MI) | · | · | |
| No (regular) | 118 (25.8) | 93 (20.4) | 323 (70.8) |
| Yes (Irregular) | 205 (45.0) | 23 (5.0) | 218 (29.2) |

## **Adverse event information**

#### 1. All-cause mortality

No deaths occurred during the intervention or follow-up period. The intervention was non-invasive and behavioral in nature.

#### 2. Serious adverse events

No serious adverse events were reported or observed. Participants were university students who voluntarily enrolled after providing informed consent. The intervention consisted of a non-invasive BCC module focused on menstrual health education. Given the educational nature and low-risk profile of the study population, no medical or psychological harm was expected or detected.

#### 3. Other (non-serious) adverse events

No non-serious adverse events exceeding the 5% frequency threshold were reported. Participants were monitored regularly throughout the study.

#### Time frame

Adverse events were monitored throughout the 6-month follow-up phase of the intervention.

## Adverse event reporting description

Adverse events were not estimated due to the non-invasive nature of the behavioral intervention.

No events were observed or self-reported during the periods of follow-up or impact assessment.

## Collection approach for table default

#### **Non-Systematic Assessment**

Adverse events were self-reported if any occurred, but no systematic daily assessment was employed.

## **Group information**

#### **Group title**

- 1. Intervention Group (participants who received BCC intervention)
- 2. Control Group (Participant s who did not received BCC intervention)

#### **Group description**

The intervention group attended BCC sessions on menstrual health, diet, and physical activity from May to June 2023, with bi-monthly follow-ups through January 2024. The control group did not receive any educational intervention. The dysmenorrhea outcome analysis included 234 participants from the intervention group and 238 from the control group. In the case of PMS and MI, 228 participants with complete and valid data were analyzed per group. To ensure baseline comparability, final analyses included 98 matched participants per group (n=196) after propensity score matching.

#### Total number affected by all-cause mortality

 Not applicable as the participants received the non-invasive nature of the behavioral intervention.

## Total number at risk for all-cause mortality

 Not applicable as the participants received the non-invasive nature of the behavioral intervention.

#### Total number at risk for serious adverse events

 Not applicable as the participants received the non-invasive nature of the behavioral intervention.

## Total number affected by any serious adverse event

 Not applicable as the participants received the non-invasive nature of the behavioral intervention. **Limitation and caveats** 

This quasi-experimental study lacked randomization, which may have introduced residual

confounding and limited causal inference. About 4% of intervention participants missed sessions

or follow-up, possibly underestimating the true effect. While the study aimed to reflect real-world

settings by conducting sessions in academic institutions, potential confounding factors related to

control group characteristics were not assessed. Dietary intake quantity was not measured, and 24-

hour recalls may have been impacted by recall bias, affecting data accuracy.

**Certain Agreements** 

Are all PIs employees of sponsor?

Yes: The principal investigator (PI) is an employee of the sponsor

There were no agreements restricting the principal investigators from discussing, presenting or

publishing the study results. The study was self-financed without external sponsorship.

**Results point of contact** 

Name or official title: Professor Dr. GM Rabiul Islam, principal investigator (PI) of the study

**Organization name:** Shahjalal University of Science and Technology, Sylhet, Bangladesh

**Phone:** +8801787323944

**Email:** rabiat14@yahoo.com

28

## References

- 1. Rupe ER, Rodean J, Hurley EA, Miller MK, Boncoeur MD, Masonbrink AR. Menstrual health among adolescents and young adults in rural Haiti. Reproductive Health. 2022;19(1):227. doi: 10.1186/s12978-022-01533-4.
- 2. Slap GB. Menstrual disorders in adolescence. Best Pract Res Clin Obstet Gynaecol. 2003;17(1):75-92. doi: https://doi.org/10.1053/ybeog.2002.0342. PubMed PMID: 12758227; PubMed Central PMCID: PMC12758227.
- 3. Sen LC, Jahan I, Salekin N, Shourove JH, Rahman M, Uddin MJ, et al. Food craving, vitamin A, and menstrual disorders: A comprehensive study on university female students. PloS one. 2024;19(9):e0310995. doi: 10.1371/journal.pone.0310995 PubMed Central PMCID: PMCPMC11423980
- 4. Andersch B, Milsom I. An epidemiologic study of young women with dysmenorrhea. American journal of obstetrics and gynecology. 1982;144(6):655-60. Epub 1982/11/15. doi: https://doi.org/10.1016/0002-9378(82)90433-1. PubMed PMID: 7137249.
- 5. Steiner M, Macdougall M, Brown E. The premenstrual symptoms screening tool (PSST) for clinicians. Archives of women's mental health. 2003;6(3):203-9. Epub 2003/08/16. doi: 10.1007/s00737-003-0018-4. PubMed PMID: 12920618.
- 6. Ansong E, Arhin SK, Cai Y, Xu X, Wu X. Menstrual characteristics, disorders and associated risk factors among female international students in Zhejiang Province, China: a cross-sectional survey. BMC women's health. 2019;19:1-10.
- 7. Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. 2020;54(24):1451-62. doi: 10.1136/bjsports-2020-102955. PubMed PMID: 33239350.

- 8. WHO. Appropriate body-mass index for Asian populations and its implications for policy and intervention strategies. Lancet (London, England). 2004;363(9403):157-63. Epub 2004/01/17. doi: 10.1016/s0140-6736(03)15268-3. PubMed PMID: 14726171.
- 9. Hanley-Cook GT, Tung JYA, Sattamini IF. Minimum Dietary Diversity for Women of Reproductive Age (MDD-W) Data Collection: Validity of the List-Based and Open Recall Methods as Compared to Weighed Food Record. 2020;12(7). doi: 10.3390/nu12072039. PubMed PMID: 32659995.
- 10. Matsuura Y, Inoue A, Kidani M, Yasui T. Change in appetite and food craving during menstrual cycle in young students. International Journal of Nutrition and Metabolism. 2020;12(2):25-30. doi: https://doi.org/10.5897/IJNAM2019.0264.
- 11. Mitsuhashi R, Sawai A, Kiyohara K, Shiraki H, Nakata Y. Factors associated with the prevalence and severity of menstrual-related symptoms: A systematic review and meta-analysis. International Journal of Environmental Research and Public Health. 2022;20(1):569.

# **Statistical Analysis Plan (SAP)**

# Statistical analysis overview

Statistical analyses were conducted to evaluate the impact of the BCC intervention on three binary outcomes: dysmenorrhea, PMS, and IMC. Categorical variables were summarized as frequencies and percentages and analyzed using the chi-square ( $\chi^2$ ) test. Continuous variables were presented as means with standard deviations and compared using independent t-tests. To adjust for potential baseline imbalances between the intervention and control groups, propensity score matching (PSM) was carried out using logistic regression. A 1:1 nearest-neighbor matching algorithm was applied with a caliper width of 0.01 and without replacement. Post-matching covariate balance was assessed using standardized mean differences (with a bias threshold of <10%) and chi-square tests. The primary analysis of intervention effects was conducted using conditional logistic regression on the matched sample. To validate the findings, bivariate and multivariate logistic regression analyses were also performed on the unmatched dataset. Additionally, sensitivity analyses were conducted to ensure the robustness and consistency of the results, including covariate balance diagnostics, estimation of the average treatment effect (ATE) and the average treatment effect on the treated (ATT), and Bayesian logistic regression on the matched sample.

# **Comparison group selection**

- 1. Intervention Group (received BCC module)
- 2. Control Group (did not receive BCC module)

**Type of statistical test:** Superiority

• Comments: The analyses were designed to assess whether the BCC intervention group had

superior outcomes compared to the control group using fixed-effect models on matched

pairs. Power calculations were based on expected reductions in outcome prevalence.

**Statistical test of hypothesis** 

Conditional logistic regression was used to estimate the odds of binary outcomes between

intervention and control groups after matching.

• P-Value: < 0.05

• Comments (P-Value): A p-value < 0.05 was considered statistically significant. No

adjustments for multiple comparisons were made. Results were considered statistically

significant at p < 0.05.

• Method: Chi-squared, t-test, regression (logistic), conditional logistic regression

• Comments (Method): Pre- and post-PSM tests used Pearson's chi-square; conditional

logistic regression applied to matched data; bivariate and multivariate logistic regression

used for robustness checks

**Method of Estimation** 

• Estimation Parameter: Odds Ratio (OR)

• Estimated Values: Reported as crude odds ratios (COR) and adjusted odds ratios (AOR).

Coefficient value was used to estimate ATE and ATT (Table 11).

• Confidence Interval Level: 95%

• Number of Sides: 2-sided

• Lower and upper limit: Reported per outcome (see Table 11)

32

- Parameter Dispersion Type: Standard error of the mean
- Estimation Comments: Odds ratios compared the intervention group (numerator) to the
  control group (reference) for menstrual outcomes. Odds ratios reflect the likelihood of
  menstrual outcomes in the intervention group relative to the control group. ATE and ATT
  were also estimated using PSM.

Table 11. Estimated odds ratios from bivariate and multivariable (before matching) as well as conditional (after matching) and logistic regression models assessing the impact of the BCC module on menstrual health outcomes

| Outcomes | Before 1 | After matching | |
|---|---|---|---|
| | COR (95% CI) | AOR (95% CI) | AOR (95% CI) |
| Dysmenorrhea | 0.07 (0.04, 0.11)*** | 0.13 (0.06, 0.26)*** | 0.13 (0.05, 0.34)*** |
| Premenstrual syndrome | 0.07 (0.04, 0.11)*** | 0.13 (0.07, 0.23)*** | 0.12 (0.06, 0.27)*** |
| Menstrual Irregularity | 0.12 (0.07, 0.20)*** | 0.26 (0.14, 0.48)*** | 0.21 (0.09, 0.45)*** |

<sup>\*</sup> Indicated chi square value define the level of significance i.e. \* p < 0.05, \*\* p < 0.01, \*\*\* p < 0.001

# Other statistical analysis

Additional scientifically appropriate analyses were conducted to ensure robustness and validity of the findings:

1. Propensity Score Matching (PSM): PSM was used to control for baseline differences between the intervention and control groups. Participants were matched 1:1 using nearest-neighbor matching with a caliper width of 0.01 and without replacement. Covariate balance was assessed using standardized mean differences (bias <10%) and post-matching chi-square tests.

- 2. Sensitivity Analyses: To confirm the quality of matching and reduce potential bias, covariate balance diagnostics were conducted, including checks for percentage bias (<10%), variance ratios (acceptable range: 0.5–2.0), and visual inspection via kernel density plots to ensure common support. Bayesian logistic regression was also applied to estimate the Log Bayes Factor, comparing models with and without the intervention to assess the strength and consistency of effects.
- **3. Alternative Estimates of Treatment Effect**: In addition to logistic regression models, the ATE an ATT were calculated (Table 12). These estimates served as supplementary measures and supported the stability of intervention effects across multiple analytical approaches.

Table 12. Estimated treatment effect of the BCC intervention on menstrual health outcomes via propensity score matching technique

| Outcomes | Average treatment effect (ATE) | | | atment effect<br>reated (ATT) |
|---|---|---|---|---|
| | Coefficient<br>(95% CI) | p-value | Coefficient<br>(95% CI) | p-value |
| Dysmenorrhea | -0.23 (-0.35, -0.11) | p < 0.001*** | -0.27 (-0.40, -0.13) | p < 0.001*** |
| Premenstrual syndrome (PMS) | -0.39 (-0.52, -0.25) | p < 0.001*** | -0.42 (-0.57, -0.26) | p < 0.001*** |
| Menstrual irregularity (MI) | -0.30 (-0.41, -0.18) | p < 0.001*** | -0.31 (-0.45, -0.16) | p < 0.001*** |

<sup>\*</sup> Indicated chi square value define the level of significance i.e. \* p < 0.05, \*\* p < 0.01, \*\*\* p < 0.001

# **Informed Consent Form (ICF)**

**Research project title:** Behavioral change communication intervention in menstrual disorder management among female university students in Bangladesh

**Objective of the study:** to evaluate the effectiveness of a structured behavior change communication intervention designed to improve menstrual health among female university students in Bangladesh.

(The interviewer will introduce herself and take consent of the interviewee before commencing the session)

#### **Introductory statement**

My name is....... I am currently working for Mr. Liton Chandra Sen, Associate Professor at the Faculty of Nutrition and Food Science, Patuakhali Science and Technology University. I have been assigned as an interviewer for the aforementioned PhD project, conducted under the Department of Food Engineering and Tea Technology at Shahjalal University of Science and Technology. Therefore, I kindly request your permission to conduct the interview, which typically takes about 15–20 minutes. We assure you that your identity will not be disclosed in any reports derived from this interview. Your confidentiality will be strictly maintained. You may skip any question or stop the interview at any time. With your consent, I would like to take written notes during the interview.

#### What will you need to do if you agree to participate?

As a selected respondent, your valuable input on a few key issues is requested. If any question makes you feel uncomfortable, you are free to skip it or not respond.

#### Risks, Benefits, confidentiality and compensation for participating

There are no risks to participating. Your input will support Mr. Sen's PhD research and help improve national reproductive health programs for young adults. All information will remain strictly confidential and used only for research by authorized personnel. Your participation in this study is completely voluntary and offers no financial compensation. There is no pressure or obligation to take part.

#### Right to refuse or withdraw

This study has been approved by the Ethical Approval Committee at Shahjalal University of Science and Technology. Participation is voluntary, and you can skip questions or withdraw at any time.

#### Who do I contact if I have a question or problem?

If you wish to know more about your rights as a participant in this study you may write Mr. Liton Chadra Sen, Associate Professor, Department of Community Health and Hygiene, Patuakhali Science and Technology University, Dumki, patuakhali-8602, email- liton.sen@pstu.ac.bd, mobile no. +8801717504808. If you have further questions regarding the nature of this study you may also contact Professor Dr. G.M. Rabiul Islam, Department of Food Engineering and Tea Technology, Shahajalal University of Science and Technology, Sylhet, email-rabiat14@yahoo.com, phone: 880 821 713 850 extn.242 (office); Cell: +88 01787323944.

#### Do you have any questions about the interview?

May we begin now? If so, please read and sign the consent form, and keep a copy for your records.

#### **Consent to publication**

This is to state that I give my full permission for the publication, reproduction, broadcast and other use of identifiable details, which can include case history and/or details within the questionnaires to be published in any Journal and Article. I confirm that I have seen and been given the opportunity to read the methodology to be published by any journal.

I understand that the published article may be available in both print and on the internet, and will be available to a broader audience through marketing channels and other third parties. Therefore, anyone can read material published in the Journal. I understand that readers may include not only public health professionals and scholarly researchers but also journalists and general members of the public. I also understand that the information will be published without my personal details and every attempt will be made to ensure anonymity.

I declare, in consequence of granting this permission, that I have no claim on ground of breach of confidence or any other ground in any legal system against the authors and its agents, publishers, successors and assigns in respect of such use of the collected information.

| Participant's Name: | Signature | Date: |
|---|---|---|
| Name of person obtaining consent: | Signature: l | Date: |
| (Individual who has been designated to obtain consent) | | |
| | | C.1 |

To be counter-signed and dated electronically for telephone interviews or in the presence of the participant for face to face interviews.